CLINICAL TRIAL: NCT00828711
Title: A Multicenter, Randomized, Double-Blind, Dose-Ranging, Phase II Study to Assess the Efficacy and Safety of the 100, 150 and 200 mcg Misoprostol Vaginal Insert for Women Requiring Cervical Ripening and Induction of Labor
Brief Title: Misoprostol Vaginal Insert (MVI) 100, 150, 200 mcg for Cervical Ripening and Induction of Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Miso-Obs-204
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Cervical Ripening; Induction of Labor
Keywords: Misoprostol vaginal insert; Induction of labor; Cervical ripening; Rate of cesarean section

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MVI 100 (Experimental): MVI 100 mcg vaginal insert
  Interventions: Drug: MVI 100
- MVI 150 (Experimental): MVI 150 mcg vaginal insert
  Interventions: Drug: MVI 150
- MVI 200 (Experimental): MVI 200 mcg vaginal insert
  Interventions: Drug: MVI 200

INTERVENTIONS:
Drug: MVI 100 — Dose reservoir of 100 mcg of misoprostol in a hydrogel polymer vaginal insert within a retrieval system. The MVI 100 will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
  Other Names: Misopess (TM); Misodel (R)
  Arms: MVI 100
Drug: MVI 150 — Dose reservoir of 150 mcg of misoprostol in a hydrogel polymer vaginal insert within a retrieval system. The MVI 150 will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
  Other Names: Misopess (TM); Misodel (R)
  Arms: MVI 150
Drug: MVI 200 — Dose reservoir of 200 mcg of misoprostol in a hydrogel polymer vaginal insert within a retrieval system. The MVI 200 will be kept in place for up to 24 hours or will be removed earlier if one of the following occur: onset of active labor, intrapartum adverse event necessitating discontinuation of the study drug, other reasons including maternal request.
  Other Names: Misopess (TM); Misodel (R)
  Arms: MVI 200

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the 100, 150 and 200 mcg Misoprostol Vaginal Insert (MVI 100, MVI 150 and MVI 200) for women requiring cervical ripening and induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Pregnant women at ≥ 36 weeks 0 days inclusive gestation;
* Women aged 18 years or older;
* Candidate for pharmacologic induction of labor;
* Single, live vertex fetus;
* Baseline modified Bishop score ≤ 4;
* Parity ≤ 3 (parity is defined as one or more births live or dead after 24 weeks gestation);
* Body Mass Index (BMI) ≤ 50 at the time of entry to the study.

Exclusion Criteria:

* Nulliparous women participating in the pharmacokinetic (PK) arm of the study: women with hemoglobin level < 11.0 grams per deciliter (g/dL) (confirmed within one week of study drug insertion);
* Women in active labor;
* Presence of uterine or cervical scar or uterine abnormality e.g., bicornate uterus. Biopsies, including cone biopsy of the cervix, are permitted;
* Administration of oxytocin or any cervical ripening or labor inducing agents (including mechanical methods) or a tocolytic drug within 7 days prior to enrollment. Magnesium sulfate is permitted if prescribed as treatment for pre-eclampsia or gestational hypertension;
* Severe pre-eclampsia marked by Hemolytic anemia, Elevated Liver enzymes, Low Platelet count (HELLP) syndrome, other end-organ affliction or Central Nervous System (CNS) findings other than mild headache;
* Fetal malpresentation;
* Diagnosed fetal abnormalities;
* Any evidence of fetal compromise at baseline (e.g., non-reassuring fetal heart rate pattern or meconium staining);
* Ruptured membranes ≥ 48 hours prior to the start of treatment;
* Suspected chorioamnionitis;
* Fever (oral or aural temperature > 37.5˚C);
* Any condition in which vaginal delivery is contraindicated e.g., placenta previa or any unexplained genital bleeding at any time after 24 weeks during this pregnancy;
* Known or suspected allergy to misoprostol, other prostaglandins or any of the excipients;
* Any condition urgently requiring delivery;
* Unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (11):
- United States (11):
  - Precision Trials, Phoenix, Arizona
  - Tuscon Medical Center, Tucson, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - UCI Medical Center, Orange, California
  - University of New Mexico Medical Center, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - University of Tennesse Medical Center, Knoxville, Tennessee
  - University of Texas Health Sciences Center at Houston, Houston, Texas

REFERENCES:
- [Derived] Wing DA, Miller H, Parker L, Powers BL, Rayburn WF; Misoprostol Vaginal Insert Miso-Obs-204 Investigators. Misoprostol vaginal insert for successful labor induction: a randomized controlled trial. Obstet Gynecol. 2011 Mar;117(3):533-541. doi: 10.1097/AOG.0b013e318209d669. PMID 21343755

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women who required to be induced were recruited at 11 sites in the US
Period: Overall Study
Arm/Group | MVI 100 | MVI 150 | MVI 200
Started | 118 | 125 | 131
Completed | 117 | 125 | 131
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVI 100 | MVI 150 | MVI 200 | Total
Number analyzed (Participants) | 117 | 125 | 131 | 373
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 117 | 125 | 131 | 373
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (6.24) | 25.8 (5.92) | 25.5 (5.93) | 25.8 (6.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 125 | 131 | 373
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 117 | 125 | 131 | 373

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women Delivering Vaginally
Time Frame: Interval from study drug administration to 24 hours
Population: Analysis based on Modified Intention-to-Treat (MITT) population who delivered vaginally. Percentage of subjects who delivered vaginally is presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 80 | 87 | 100
percentage of participants | 63.75 [52.24 to 74.21] | 66.67 [55.75 to 76.42] | 76.00 [66.43 to 83.98]
Statistical Analysis 1: Comparison: MVI 100 vs MVI 200; The primary objective of this study is to compare the efficacy of MVI 100 and MVI 200 based on the proportion of vaginal deliveries within 24 hours. A minimum sample size of approximately 120 subjects per arm would provide 84 subjects per arm with vaginal delivery, which would ensure >80% power (with two-sided alpha of 5%) to detect a 20% improvement in the proportion of women delivering vaginally within 24 hours; Test type: Superiority or Other; p = 0.057, Cochran-Mantel-Haenszel; Adjusted for site effect; Difference in Proportions = 12.20 — MVI 200 - MVI 100

2. Secondary Outcome: Time to Vaginal Delivery
Time Frame: Interval from study drug administration to delivery (average 24 hours)
Population: Kaplan-Meier Estimates are based on Modified Intention-to-Treat (MITT) population.Subjects who had a cesarean, discharged prior to delivery or withdrew consent during first hospitalization were censored (MVI 100: 37, MVI 150: 39, MVI 200: 31) using the longest time interval from study drug administration to cesarean or to Labor & Delivery discharge
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 117 | 125 | 131
minutes | 1744 [1368 to 2198] | 1535 [1292 to 2063] | 1181 [1035 to 1443]
Statistical Analysis 1: Comparison: MVI 100 vs MVI 200; Subjects who underwent a cesarean delivery during the first hospitalization were censored using the longest time interval from study drug administration to cesarean delivery during the first hospitalization, independent of treatment group. Subjects who, in their first hospitalization, were discharged prior to delivery or withdrew consent prior to delivery were censored using the longest time interval from study drug administration to labor and delivery discharge, independent of treatment group; Test type: Superiority or Other; p = 0.018, Log Rank; Median Difference (Net) = -563 — MVI 200 - MVI 100

3. Secondary Outcome: Rate of Adverse Events
Description: All adverse events were rated by the Investigator as mild, moderate or severe and classified as having no relationship, possible relationship or a probable relationship to the study drug. These assessments were deemed as accurate and appropriate for the reporting of all serious and non serious adverse events.
Time Frame: From study drug administration to hospital discharge (approximately 48 - 72 hours)
Population: The percentage of subjects with adverse events are presented for the Intrapartum (before delivery), postpartum (maternal) and neonatal periods.
Measure: Number; unit: percentage of participants
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 118 | 125 | 131
percentage of participants
  Subjects with Intrapartum Adverse Events | 81.4 | 80.0 | 79.4
  Subjects with Maternal Postpartum Adverse Events | 28.0 | 27.2 | 32.1
  Subjects with Neonatal Adverse Events | 39.8 | 42.4 | 48.9

4. Secondary Outcome: Proportion of Cesarean Delivery
Time Frame: Interval from study drug administration to cesarean delivery (average 24 hours)
Population: Percentage of subjects who had a cesarean delivery during the first hospitalization (safety population) is presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 118 | 125 | 131
percentage of participants | 31.36 [23.13 to 40.54] | 30.40 [22.49 to 39.26] | 22.90 [16.02 to 31.05]
Statistical Analysis 1: Comparison: MVI 100 vs MVI 200; Test type: Superiority or Other; p = 0.153, Fisher Exact; Difference in Proportions = -8.46 — MVI 200 - MVI 100

5. Secondary Outcome: Cervical Ripening Using Composite Measure of Success
Description: Cervical ripening success was defined by achievement of one or more of the following by 12 hours after study drug administration:
  * Increase from baseline in modified Bishop score ≥3; or
  * Achievement of modified Bishop score of ≥6; or
  * Vaginal delivery.
Time Frame: 12 hours after insertion of drug
Population: Percentage of subjects with cervical ripening success at 12 hours is presented (Modified Intention-to-Treat population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 117 | 125 | 131
percentage of participants | 77.78 [69.16 to 84.94] | 77.60 [69.28 to 84.57] | 80.15 [72.29 to 86.61]
Statistical Analysis 1: Comparison: MVI 100 vs MVI 200; Test type: Superiority or Other; p = 0.65, Cochran-Mantel-Haenszel; Adjusted for site effect; Difference in Proportions = 2.37 — MVI 200 - MVI 100

6. Secondary Outcome: Use of Oxytocin
Description: Percentage of participants in receipt of Oxytocin for induction after study drug removal is accurate and appropriate for this outcome measure.
Time Frame: At least 30 minutes after study drug removal
Population: Percentage of subjects who required pre-delivery oxytocin is presented (Modified Intention-to-Treat population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 117 | 125 | 131
percentage of participants | 70.94 [61.83 to 78.96] | 60.00 [50.86 to 68.66] | 48.85 [40.03 to 57.74]
Statistical Analysis 1: Comparison: MVI 100 vs MVI 200; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel; Adjusted for site effect; Difference in Proportions = -22.09 — MVI 200 - MVI 100

7. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax), Maximum Plasma Concentration (Cmax), Area Under the Curve (AUC) and Terminal Half Life of Misoprostol Acid.
Description: The timepoints over which the pharmacokinetic measurements were assessed, and deemed as accurate and appropriate, were as follows: 0 hours (baseline), 2, 4, 6, 8, 10 and 14 hours after insertion of the study drug, immediately prior to removal of the study drug and 0.5, 1 and 2 hours after removal of the study drug.
Time Frame: From study drug insertion up to 2 hours post study drug removal
Population: The plan was to enrol 24 subjects to the pharmacokinetic (PK) arm of the study. Only 3 subjects enrolled in the PK arm; there were too few subjects and too few samples available. Due to insufficient data, no statistical analysis was possible. Only misoprostol acid levels for each blood sampling timepoint for each subject was determined.
Measure: Number; unit: PK Parameters
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 1 | 2 | 0
PK Parameters | NA — Only misoprostol acid levels for each blood sampling timepoint for this one subject was determined. Due to insufficient data no statistical analysis of PK parameters was possible. | NA — Only misoprostol acid levels for each blood sampling timepoint for these two subjects were determined. Due to insufficient data no statistical analysis of PK parameters was possible. |

8. Secondary Outcome: Time to Onset of Active Labor
Time Frame: Interval from study drug administration to active labor (average 12 hours)
Population: Kaplan-Meier Estimates for Time to Onset of Active Labor presented (Modified Intention-to-Treat population). Subjects who never went into active labor during the first hospitalization were censored using the longest time interval from study drug administration to delivery (Censored subjects = MVI 100: 5; MVI 150: 7; MVI 200: 8)
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | MVI 100 | MVI 150 | MVI 200
Number analyzed (Participants) | 117 | 125 | 131
minutes | 1069.00 [885.0 to 1153.0] | 775.00 [724.0 to 977.0] | 701.00 [550.0 to 759.0]
Statistical Analysis 1: Comparison: MVI 100 vs MVI 200; Subjects who never went into active labor during the first hospitalization were censored using the longest time interval from study drug administration to delivery during the first hospitalization, independent of treatment group. Subjects who, in their first hospitalization, were discharged prior to delivery or withdraw consent prior to delivery will be censored using the longest time interval from study drug administration to labor and delivery discharge, independent of treatment group; Test type: Superiority or Other; p = 0.007, Log Rank; Median Difference (Net) = -368 — MVI 200 - MVI 100

ADVERSE EVENTS:
Time Frame: All adverse events were followed until resolution or for at least 30 days after discontinuation of study drug, whichever occurred first.
Description: All adverse events occurring to the maternal-fetal unit (pre-delivery/ intrapartum), the mother (postpartum) or the neonate were recorded. Adverse events that resulted in a cesarean delivery were reported as serious adverse events as they were medically significant events that routinely prolonged the duration of hospitalization.
Arm/Group | MVI 100 | MVI 150 | MVI 200
Serious Adverse Events (participants affected / at risk) | 43/118 | 48/125 | 42/131
Other Adverse Events (participants affected / at risk) | 100/118 | 107/125 | 117/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVI 100 (N=118) | MVI 150 (N=125) | MVI 200 (N=131)
Ankyloglossia congenital * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Atrial septal defect * (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) — * Neonatal Event
Dysmorphism * (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) — * Neonatal Event
Polydactyly * (Congenital, familial and genetic disorders) | 0 (0) | 3 (3) | 5 (5) — * Neonatal Event
Supernumerary nipple * (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) — * Neonatal Event
Syndactyly * (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Dacryostenosis congenital * (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Fever neonatal * (General disorders) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Congenital syphilis * (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — * Neonatal Event
Endometritis # (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — # Postpartum Event
Herpes simplex * (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Postoperative wound infection # (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — # Postpartum Event
Arterial injury # (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — # Postpartum Event
Post procedural haemorrhage # (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — # Postpartum Event
Medical observation * (Investigations) | 0 (0) | 0 (0) | 1 (1) — * Neonatal Event
Urine cannabinoids increased + (Investigations) | 0 (0) | 1 (1) | 0 (0) — + Intrapartum Event
Dehydration * (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — * Neonatal Event
Feeding disorder neonatal * (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) — * Neonatal Event
Haemorrhage intracranial * (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — * Neonatal Event
Hydrocephalus * (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — * Neonatal Event
Abnormal labour affecting foetus + (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — + Intrapartum Event
Arrested labour + (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 16 (16) | 11 (11) — + Intrapartum Event
Chorioamnionitis + (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) — + Intrapartum Event
Drug withdrawal syndrome neonatal + (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 2 (2) — + Intrapartum Event
Foetal heart rate disorder + (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 12 (12) | 18 (18) — + Intrapartum Event
Foetal malpresentation + (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — + Intrapartum Event
Hyperbilirubinaemia neonatal * (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 7 (7) | 6 (6) — * Neonatal Event
Hypoglycaemia neonatal * (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 2 (2) — * Neonatal Event
Neonatal disorder * (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — * Neonatal Event
Postpartum haemorrhage # (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — # Postpartum Event
Pre-eclampsia + (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — + Intrapartum Event
Pre-eclampsia # (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — # Postpartum Event
Puerperal pyrexia # (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — # Postpartum Event
Small for dates baby * (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — * Neonatal Event
Uterine cervical laceration during labour # (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — # Postpartum Event
Renal failure acute # (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — # Postpartum Event
Penis disorder * (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Vaginal haematoma # (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — # Postpartum Event
Vulval haematoma + (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — + Intrapartum Event
Neonatal hypoxia * (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — * Neonatal Event
Pulmonary oedema # (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — # Postpartum Event
Infection prophylaxis * (Surgical and medical procedures) | 2 (2) | 2 (2) | 0 (0) — * Neonatal Event
Hypertension # (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — # Postpartum Event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVI 100 (N=118) | MVI 150 (N=125) | MVI 200 (N=131)
Anaemia # (Blood and lymphatic system disorders) | 10 (10) | 8 (8) | 11 (11) — # Postpartum Event
Abnormal labour affecting foetus + (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 12 (14) | 16 (16) — + Intrapartum Event
Caput succedaneum * (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 5 (5) | 7 (7) — * Neonatal Event
Chorioamnionitis + (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 7 (7) | 2 (2) — + Intrapartum Event
Foetal heart rate disorder + (Pregnancy, puerperium and perinatal conditions) | 67 (96) | 62 (79) | 57 (87) — + Intrapartum Event
Hyperbilirubinaemia neonatal * (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 6 (6) | 10 (10) — * Neonatal Event
Meconium in amniotic fluid + (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 13 (13) | 22 (22) — + Intrapartum Event
Postpartum haemorrhage # (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 5 (5) | 8 (8) — # Postpartum Event
Umbilical cord around neck * (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 11 (11) | 22 (22) — * Neonatal Event
Uterine contractions abnormal + (Pregnancy, puerperium and perinatal conditions) | 23 (23) | 32 (33) | 54 (57) — + Intrapartum Event
Uterine hypertonus + (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 7 (7) | 9 (9) — + Intrapartum Event
Uterine atony # (Reproductive system and breast disorders) | 5 (5) | 9 (9) | 6 (6) — # Postpartum Event
Neonatal respiratory distress syndrome * (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 5 (5) — * Neonatal Event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any abstract,presentation or manuscript proposed for publication must be submitted to the Sponsor for review at least 30 days prior to submission for any meeting or journal.If deemed necessary by the Sponsor for protection of proprietary information prior to patent filing,the Investigator agrees to a further delay of 60 days before any presentation or publication is submitted.Publications must be in a form that does not reveal technical information that is considered confidential or proprietary.